CLINICAL TRIAL: NCT04714463
Title: Psychological Effect of Expectations and Body Image on Outcomes of Breast Reconstruction
Brief Title: Effects of Expectations and Body Image in Breast Reconstruction
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020-06245
Record Dates: First submitted 2021-01-12; First posted 2021-01-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: plastic surgery; breast reconstruction; complication; expectations; body image
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immediate breast reconstruction: Women undergoing immediate breast reconstruction due to breast cancer or a high risk for breast cancer
  Interventions: Procedure: Implant-based breast reconstruction; Procedure: Autologous breast reconstruction; Procedure: Combined methods
- Delayed breast reconstruction: Women undergoing delayed breast reconstruction due to breast cancer or a high risk for breast cancer
  Interventions: Procedure: Implant-based breast reconstruction; Procedure: Autologous breast reconstruction; Procedure: Combined methods

INTERVENTIONS:
Procedure: Implant-based breast reconstruction — All types of implant based breast reconstructions
Procedure: Autologous breast reconstruction — All types of autologous breast reconstructions
Procedure: Combined methods — All types of breast reconstructions combining autologous and implant based techniques

SUMMARY:
A breast reconstruction after mastectomy, either due to breast cancer or a high lifetime risk for cancer, is performed to increase the patient's quality of life. However, there are studies that show that some women regret their decision to have breast reconstruction. There are also studies demonstrating similarities in the general patterns of psychosocial adjustment and quality of life among women with breast cancer who have undergone breast-conserving surgery, mastectomy alone, and mastectomy combined with breast reconstruction. Hence, it is unclear which women actually beneﬁt from a breast reconstruction. The concept of quality of life is connected to patient satisfaction and body image/investment. Therefore, the aim of this project is to examine the effects of patient expectations and body image on the patient reported outcomes of breast reconstruction, to improve preoperative information and postoperative care for women considering a breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Biological women with breast cancer or high risk for breast cancer who want post-mastectomy breast reconstruction
* Age > 18 years

Exclusion Criteria:

* Inability to give informed consent
* Inability to understand Swedish
* Relaps of cancer
* Palliative treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological women with breast cancer or high risk for breast cancer who want post-mastectomy breast reconstruction
Study Population: Biological women with breast cancer or high risk for breast cancer who want immediate or delayed post-mastectomy breast reconstruction.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction with breast reconstruction measured with Breast Q reconstruction | 2 years
  Breast Q reconstruction includes two domains and six different modules: health-related quality of life (HR-QOL; including physical, psychosocial, and sexual well-being) and patient satisfaction (including satisfaction with breasts, outcome, and care). Each scale produces an independent score from 0-100. A higher score means greater satisfaction or better QOL.
Patient expectations measured with Breast Q expectations | 2 years
  Breast Q expectations.The scale consists of five modules: expectations for support from medical staff , expectations for pain, expectations for coping, expectations for breast appearance when clothed and expectations for breast sensation. The score for each independent scale range from 0-100. A higher score means greater expectations.
Body image measured with Multidimensional body-self relations questionnaire- appearance scales (MBSRQ-AS) | 2 years
  MBSRQ-AS - Multidimensional body-self relations questionnaire- appearance scales.It is a 34-item self-report questionnaire designed to measure appearance related components of body-image. In consists of five subscales: appearance evaluation, appearance orientation, body areas satisfaction, overweight preoccupation, and self-classified weight. It is a 5-point Likert-scale ranging from 1 to 5.
Body image investment measured with Appearance schemas inventory-revised (ASI-R) | 2 years
  ASI-R - Appearance schemas inventory-revised: is a 20-item self-report questionnaire designed to measure body-image investment. It consists of two subscales, self-evaluative salience (SES) and motivational salience (MS). It is a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). Twelve items relate to SES and eight items relate to MS. The total score is the mean of the 20 items, and the score of the subscales is the mean of the items relating to each subscale. A high score indicates greater body-image investment.

SECONDARY OUTCOMES:
Satisfaction with preoperative information measured with Breast Q reconstruction | 2 years
  Measured with one of the sub scales of Breast Q reconstruction
Pain measured with a visual analogue scale | 2 weeks
  Measured with a post-operative pain dairy with VAS scales (o means no pain and 10 means the worst possible pain imaginable)
Sick leave according to authorities | 1 year
  Actual sick leave according to the Swedish authorities
Number of out-patient visits according to the medical charts | 1 year
  Actual number of out-patient visits, according to the medical chart
Depression and anxiety measured with Hospital Anxiety and Depression Scale (HADS) | 2 years
  HADS - Hospital Anxiety and Depression Scale: is a 14-item self-report questionnaire that is designed to measure anxiety and depression. It has two domains, where seven items relate to anxiety and seven relate to depression. It is a 4-point Likert-scale ranging from 0-3. Each domain has a maximum score of 21. For both domains, scores of less than 7 indicate non-cases, whereas scores of 8-10 indicate mild anxiety or depression, 11-14 moderate and 15-21 severe.
Demographic factors and medical factors according to medical charts | 2 years
  Demographic factors that might affect expectations and satisfaction, such as age, comorbidity, and previous cosmetic breast surgery, and medical factors such as timing of reconstructions, reason for mastectomy, type of cancer and cancer treatment received.

OTHER OUTCOMES:
Translation and validation of Breast-Q expectations | 4 months
  Translation into Swedish according to MAPI-guidelines. Validation of psychometric properties in a Swedish population.The scale consists of five modules: expectations for support from medical staff , expectations for pain, expectations for coping, expectations for breast appearance when clothed and expectations for breast sensation. The score for each independent scale range from 0-100. A higher score means greater expectations.
Translation and validation of Appearance schemas inventory-revised (ASI-R) | 4 months
  Translation into Swedish according to MAPI-guidelines. Validation of psychometric properties in a Swedish population. ASI-Ris a 20-item self-report questionnaire designed to measure body-image investment. It consists of two subscales, self-evaluative salience (SES) and motivational salience (MS). It is a 5-point Likert-scale ranging from 1 (strongly disagree) to 5 (strongly agree). Twelve items relate to SES and eight items relate to MS. The total score is the mean of the 20 items, and the score of the subscales is the mean of the items relating to each subscale. A high score indicates greater body-image investment.
Translation and validation of Multidimensional body-self relations questionnaire- appearance scales (MBSRQ-AS) | 4 months
  Translation into Swedish according to MAPI-guidelines. Validation of psychometric properties in a Swedish population.Multidimensional body-self relations questionnaire- appearance scales.It is a 34-item self-report questionnaire designed to measure appearance related components of body-image. In consists of five subscales: appearance evaluation, appearance orientation, body areas satisfaction, overweight preoccupation, and self-classified weight. It is a 5-point Likert-scale ranging from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hansson, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jepsen C, Paganini A, Hansson E. Validation and reliability testing of the Swedish version of the BREAST-Q reconstruction. Scand J Surg. 2025 Oct 26:14574969251387498. doi: 10.1177/14574969251387498. Online ahead of print. PMID 41139858
- [Derived] Weick L, Grimby-Ekman A, Lunde C, Hansson E. Validation and reliability testing of the BREAST-Q expectations questionnaire in Swedish. J Plast Surg Hand Surg. 2023 Feb-Dec;57(1-6):315-323. doi: 10.1080/2000656X.2022.2070180. Epub 2022 May 9. PMID 35533094